CLINICAL TRIAL: NCT02986776
Title: Treatment Settings for Alcoholics: A Field Extension
Brief Title: Treatment Settings for Those With an Alcohol Problem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Rychtarik, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA013625
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Abuse; Alcohol-dependence
MeSH Terms: conditions — Alcoholism | interventions — Hospitalization; Ambulatory Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Inpatient Care + Needs Inpatient (Active Comparator): Individuals with high alcohol involvement or low cognitive functioning receiving inpatient treatment
  Interventions: Behavioral: Inpatient Care
- Inpatient Care + No Need for Inpatient (Active Comparator): Individuals with low alcohol involvement or mid-high cognitive functioning receiving inpatient treatment
  Interventions: Behavioral: Inpatient Care
- Outpatient Care + Needs Inpatient (Active Comparator): Individuals with high alcohol involvement or low cognitive functioning receiving outpatient treatment
  Interventions: Behavioral: Outpatient Care
- Outpatient Care + No Need for Inpatient (Active Comparator): Individuals with low alcohol involvement and or mid-high cognitive functioning receiving outpatient treatment
  Interventions: Behavioral: Outpatient Care

INTERVENTIONS:
Behavioral: Inpatient Care — 21 days of inpatient substance misuse treatment
  Arms: Inpatient Care + Needs Inpatient; Inpatient Care + No Need for Inpatient
Behavioral: Outpatient Care — 21 days of outpatient substance misuse treatment
  Arms: Outpatient Care + Needs Inpatient; Outpatient Care + No Need for Inpatient

SUMMARY:
A prior study in a tightly controlled clinical research environment found individuals with an alcohol use disorder (AUD) benefited more from inpatient (IP) than outpatient (OP) care, if they presented with high alcohol involvement and/or low cognitive functioning. This study sought to: (a) validate and extend these findings within the uncontrolled environment of a community-based treatment center, and (b) test whether inpatients had fewer days of involuntary abstinence (e.g., incarcerations) relative to outpatients. Based on their need for inpatient treatment, using prior cut-points for alcohol involvement and cognitive functioning, participants were randomly assigned within inpatient need group (No Need for IP; Needs IP) to either 21-days of inpatient substance misuse treatment or 21-days of outpatient treatment, all followed by 6 months of continuing outpatient care. Follow-up were conducted an 90-day intervals across 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for treatment through the Chemical Dependency treatment programs of a large, community-based healthcare network
* Drank alcoholic beverages within the last 90 days
* Have a current address (not homeless)
* Free of legal stipulations that would affect treatment decisions
* Have a past 3 months Alcohol Use Disorder
* Primary alcohol, or alcohol and drug problem

Exclusion Criteria:

* Homeless
* Drug problem only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2002-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Monthly Percentage of Voluntary Abstinent Days (from Timeline Followback Interview) | Change up to 18 months
  Percentage of Days Abstinent of those in which drinking was not restricted
Monthly Point Prevalence of Abstinent Days (from Timeline Followback Interview) | Change up to 18 months
  Monthly percentage of participants abstinent throughout a month
Monthly Drinks per Drinking Day (from Timeline Followback Interview) | Change up to 18 months
  For those drinking in a month, average drinks per drinking day

SECONDARY OUTCOMES:
Monthly percentage of Involuntary abstinent days (from Timeline Followback Interview) | Up to 18 months
  Monthly percentage of days in which the participant was incarcerated, hospitalized, or in residential treatment

REFERENCES:
- [Derived] Rychtarik RG, McGillicuddy NB, Papandonatos GD, Whitney RB, Connors GJ. Randomized clinical trial of matching client alcohol use disorder severity and level of cognitive functioning to treatment setting: A partial replication and extension. Psychol Addict Behav. 2017 Aug;31(5):513-523. doi: 10.1037/adb0000253. Epub 2017 Feb 2. PMID 28150955